CLINICAL TRIAL: NCT04889599
Title: An Open Label, Two Treatment, Two Period, Two Sequence,Crossover, Bioequivalence Study of BH009 Against Winthrop (Docetaxel) Injection in Patients With Solid Tumors
Brief Title: A Bioequivalence Study of Docetaxel Injection in Patients With Solid Tumours
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhuhai Beihai Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20-VIN-0225
Record Dates: First submitted 2021-04-25; First posted 2021-05-17 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-05

CONDITIONS: Docetaxel; Solid Tumours; Bioequivalence
MeSH Terms: interventions — Docetaxel; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BH009 (Docetaxel Injection) (Experimental): Patients will receive single dose BH009 75 mg/m2, as a 1-hour IV infusion.
  Interventions: Drug: BH009 (Docetaxel injection)
- Docetaxel Injection (Active Comparator): Patients will receive single dose Docetaxel Injection 75 mg/m2, as a 1-hour IV infusion.
  Interventions: Drug: Docetaxel injection

INTERVENTIONS:
Drug: BH009 (Docetaxel injection) — 75mg/m2
  Other Names: BH009
  Arms: BH009 (Docetaxel Injection)
Drug: Docetaxel injection — 75mg/m2
  Other Names: Winthrop (Docetaxel) Injection
  Arms: Docetaxel Injection

SUMMARY:
The study will be conducted in patients with solid tumors for whom single-agent docetaxel, in the dose of 75 mg/m2, is a suitable treatment option. Each patient, meeting all the inclusion criteria and none of the exclusion criteria, will receive test or reference product in a cross over manner based on randomization schedule. A balance between T-R and R-T randomization sequence will be ensured using statistical techniques. Blood samples for PK assessment will be collected prior to and after start of intravenous infusion on Day 1 (Period I), Day 22 (Period II)

DETAILED DESCRIPTION:
46 patients will be enrolled in the study.

The dosing schedule will be as follows:

Period I (Day 1): Patients will receive 75 mg/m2 dose of docetaxel injection for infusion (either test or reference product) on the first day of the chemotherapy cycle.

Period II (Day 22): Patients will be crossover to another treatment arm to receive 75 mg/m2 dose of docetaxel injection for infusion (either test or reference product depending of crossover sequence) on the first day of the next chemotherapy cycle.

A total of 17 blood samples for PK assessment will be collected during each period.

The pre-infusion blood sample of 06 mL (0.000 hr) will be collected within 5 minutes prior to start of infusion.

On Day 1 (Period I) and Day 22# (Period II):

The blood samples of 06 mL each will be drawn at 0.500 (30 minutes), 0.667 (40 minutes) and 0.833 (50 minutes) during infusion, 1.000 hour* (immediately at the actual end of infusion), and at 0.083 (5 minutes), 0.167 (10 minutes), 0.333 (20 minutes), 0.500 (30 minutes), 1.000, 2.000, 3.000, 6.000, 8.000, 12.000, 24.000 and 48.000 hours after the end of the docetaxel infusion.

Employing the estimated concentration time profiles of Unbound Docetaxel & Total Docetaxel following variables will be calculated:

Primary variables: Cmax, AUC0-t and AUC0-∞

Secondary variable: Tmax, t1/2, Kel, Vd, CL and AUC_%Extrap_obs

Criteria for evaluation:

For Unbound Docetaxel & Total Docetaxel, based on the statistical results of 90% confidence intervals for the geometric least square mean ratio (T/R) for the pharmacokinetic parameters Cmax, AUC0-t and AUC0-∞, conclusions will be drawn whether test formulation is bioequivalent to reference formulation. Acceptance range for bioequivalence is 80.00% - 125.00% for 90% confidence intervals of the geometric least square means ratio (T/R) for Cmax, AUC0-t and AUC0-∞.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all of the following criteria will be considered for enrollment in the study.

1. Patients of either gender, ≥18 years of age.
2. Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures.
3. Histologically or cytologically confirmed advanced solid tumors who are scheduled to receive treatment with single-agent docetaxel, in the dose of 75 mg/m2 or those whose are already receiving single-agent docetaxel (taxotere® or an approved generic drug of taxotere®), in the dose of 75 mg/m2 and are scheduled to two more cycles, in the same dose, as per the actual treatment plan. Note: Metastatic castration-resistant prostate cancer will not be considered for the study as the patients are required to receive prednisone along with docetaxel and the regime of dexamethasone (CYP 3A4 inducer is different from that in other indications)
4. ECOG performance status 0 or 1 and Life expectancy ≥3 months (as per the Investigator's discretion).
5. Adequate Hematopoietic, Renal and Liver function defined as the following:

   Bone marrow function :ANC ≥1500/mm3, Platelet count ≥100,000/mm3, Haemoglobin > 9.0 g/dl Hepatic function:ALT/AST ≤ 1.5 × ULN, Alkaline phosphatase ≤ 2.5 × ULN ,Total Bilirubin ≤ ULN Renal function:Serum creatinine ≤1.5 x ULN
6. Prothrombin time, international normalized ratio or activated partial thromboplastin time <1.5 × ULN; Use of full dose anticoagulants is permitted. These laboratories should be maintained within the therapeutic range and closely monitored by the Investigator.
7. Recovery, to Grade 0-1 (as per CTCAE 5.04 criteria), from adverse events related to prior anticancer therapy except alopecia and endocrinopathies controlled with hormone replacement therapy.
8. Prior chemotherapy (except ongoing taxotere or an approved generic of taxotere, in which last dose must have been received at least 21 days prior to cycle 1 of the study), immunotherapy and radiation therapy must be completed at least 30 days prior to randomization (42 days for mitomycin C or nitrosoureas). Completion of palliative radiotherapy to a single disease site must be completed at least 14 days prior to randomization.
9. In case of female patient, the serum pregnancy test at screening visit and urine pregnancy test at baseline must be negative.
10. Sexually active women, unless surgically sterile (at least 6 months prior to Study drug administration) or postmenopausal for at least 12 consecutive months, must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives [any hormonal method in conjunction with a secondary method], intrauterine device, female condom with spermicide, diaphragm with spermicide, absolute sexual abstinence, use of condom with spermicide by sexual partner or sterile [at least 6 months prior to Study drug administration] sexual partner) for at least 1 month prior to study drug administration, during study and up to 6 month after the last dose of study drug. Cessation of birth control after this point should be discussed with a responsible physician.
11. In case of male patients: either partner or patient must use an effective method of avoiding pregnancy for at least 1 month prior to study drug administration, during study and up to 3 month after the last dose of study drug. Cessation of birth control after this point should be discussed with a responsible physician.

Exclusion Criteria:

Patients will be excluded from the study, if they meet any of the following criteria:

1. Hypersensitivity or idiosyncratic reaction to docetaxel, its excipients, and/or related substances including polysorbate 80, paclitaxel, alcohol, dexamethasone and Antiemetic (Granisetron or Ondansetron).
2. Severe cardiovascular disease, including CVA, TIA, myocardial infarction, or unstable angina within 6 months of study entry; NYHA class III or IV heart failure within 6 months of study entry; uncontrolled arrhythmia within 6 months of study entry.
3. Average corrected QT (QTc) interval by Frederica's formula (QTcF) on triplicate ECGs at screening > 470 msec (females) or > 450 msec (males); or on concomitant medications that would prolong the QT interval; or have family history of long QT syndrome.
4. Patients with an active infection (e.g. tuberculosis, sepsis and opportunistic infections).
5. Patients with severe pleural effusion (volume involving > 40% of the hemithorax on CT scan chest) or gross ascites (>800ml of ascitic fluid)3,4.
6. Peripheral neuropathy ≥grade 2 (as per CTCAE 5.04 criteria).
7. A positive hepatitis screen including hepatitis B surface antigen and HCV antibodies.
8. Patients with HIV infection.
9. Patients with known brain metastasis or those showing neurologic symptoms due to brain metastasis.
10. Recent or clinically significant history of drug or alcohol abuse.
11. Patients require concomitant treatment with potent Cytochrome P450 3A4 inhibitors, inducers or substrates.
12. Use of any Cytochrome P450 3A4 inducers, inhibitors, or substrates that may alter docetaxel metabolism (e.g. dronedarone, epirubicin, sorafenib, CNS depressants) within 14 days before randomization.
13. Major surgery within 4 weeks prior to study entry; minor surgery within 2 weeks prior to study entry.
14. Patients found positive on urine scan for drugs of abuse and/or breath test for alcohol consumption at screening or baseline. Note: Benzodiazepines and /or opioids given in therapeutic doses under the observation of physician for management of insomnia / anxiety / pain, etc., will be allowed, provided that there is no drug-drug interaction with the study drug and an approval from the Veeda medical monitor is taken.
15. The receipt of an investigational medicinal product or participation in other drug research study within a period of 30 days (or 5 half-lives, whichever is longer) prior to the first dose of investigational medicinal product for the current study.
16. Pregnant or Breast feeding female.
17. Donation of blood (1 unit or 350 ml) within 90 days prior to receiving the first dose of investigational medicinal product for the current study.
18. Abnormal baseline laboratory / physical findings considered to be clinical significant by the investigator.
19. Patients with any significant history of non-compliance or inability to reliably grant informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Cmax of docetaxel injection | On Day 1 (Period I) and Day 24 (Period II)
  Peak Plasma Concentration
AUC of docetaxel injection | On Day 1 (Period I) and Day 24 (Period II)
  Area under the plasma concentration versus time curve

SECONDARY OUTCOMES:
To evaluate of safety and tolerability of BH009 | From the Period I Day 1 to 7 days after the last dose
  Adverse event assessments included laboratory test values, patient reports, and investigator observations.
  Number of participants and order of severity with treatment-related adverse events as assessed by CTCAE 5.04.

CONTACTS AND LOCATIONS:
Overall Officials: Gopichand M, Ph. D., Principal Investigator — HCG City Cancer center
Locations (3):
- India (3):
  - HCG City Cancer center, Āndra
  - Nirmal Hospital Pvt. Ltd, Gujrāt
  - HCG Manavata Cancer Centre, Mahara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho EK, Park JY, Lee KH, Song HS, Min YJ, Kim YH, Kang JH. Open-label, randomized, single-dose, crossover study to evaluate the pharmacokinetics and safety differences between two docetaxel products, CKD-810 and Taxotere injection, in patients with advanced solid cancer. Cancer Chemother Pharmacol. 2014 Jan;73(1):9-16. doi: 10.1007/s00280-013-2264-0. Epub 2013 Dec 12. PMID 24337589
- See also: Cancer Chemother Pharmacol. 2014 Jan;73(1):9-16. doi: 10.1007/s00280-013-2264-0. Epub 2013 Dec 12. — https://pubmed.ncbi.nlm.nih.gov/24337589/